CLINICAL TRIAL: NCT00749021
Title: A Phase I Study to Evaluate the Efficacy and Safety of Treating Subfoveal Pigment Epithelial Detachment Associated With Choroidal Neovascularization With Anti-vascular Endothelial Growth Factor Fragment, Ranibizumab.
Brief Title: Ranibizumab for Treating Submacular Vascularized Pigment Epithelial Detachments
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Clement K. Chan (Other)
Responsible Party: Sponsor-Investigator, Clement K. Chan, Principal Investigator, Southern California Desert Retina Consultants, MC
Organization: Southern California Desert Retina Consultants, MC (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FVF4332s
Record Dates: First submitted 2008-09-08; First posted 2008-09-09 (Estimated); Last update posted 2012-10-05 (Estimated); Status verified 2012-10

CONDITIONS: Retinal Pigment Epithelial Detachment
Keywords: choroidal neovascularization; vascularized
MeSH Terms: conditions — Retinal Detachment; Choroidal Neovascularization; Neovascularization, Pathologic | interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Regimen 1 (Active Comparator): Intravitreal injection of Ranibizumab monthly for 12 months.
  Interventions: Drug: Ranibizumab
- Regimen 2 (Active Comparator): Intravitreal injection of ranibizumab for 4 months (at Day 0, Month 1, Month 2, and Month 3) followed by by treatments on predefined re-treatment criteria.
  Interventions: Drug: Ranibizumab
- Regimen 3 (Active Comparator): Intravitreal injection of Ranibizumab 2.0mg monthly for 12 months
  Interventions: Drug: Ranibizumab
- Regimen 4 (Active Comparator): Intravitreal injection 2.0mg ranibizumab for 4 months (at Day 0, Month 1 and Month 2, and Month 3) followed by PRN treatments on pre-defined re-treatment criteria
  Interventions: Drug: Ranibizumab

INTERVENTIONS:
Drug: Ranibizumab — 0.5 mg of intravitreal ranibizumab monthly for 12 months
  Other Names: Lucentis
  Arms: Regimen 1
Drug: Ranibizumab — 0.5 mg intravitreal injection of ranibizumab for 4 months followed by PRN dosing
  Other Names: Lucentis
  Arms: Regimen 2
Drug: Ranibizumab — 2.0mg of intravitreal ranibizumab monthly for 12 months
  Other Names: Lucentis
  Arms: Regimen 3
Drug: Ranibizumab — 2.0mg of intravitreal injection of Ranibizumab for 4 months followed by PRN dosing
  Other Names: Lucentis
  Arms: Regimen 4

SUMMARY:
This is a multicenter, randomized, open-label study. 40 patients will be followed for a period of 12 months. All consented and enrolled patients will receive either 0.5mg or 2.0mg of intravitreal ranibizumab injection.

ELIGIBILITY:
Inclusion Criteria:

* Patient is 50 years or older
* Patient is willing to participate in this study and to follow the criteria and protocol of this study.
* Patient is not involved with another clinical trial.
* Ability to understand the informed consent and willingness to sign the consent.
* Presence of a submacular vascularized or fibrovascular PED. Central foveal involvement by the PED or the CNV due to age related macular degeneration.
* PED less than or equal to 12 disc area in size
* BCVA with ETDRS of greater than or equal to 19 letters and less than or equal to 69 letters (20/400 to 20/40)
* Central 1-mm foveal thickness of greater than or equal to 250 microns on OCT.
* Greatest linear diameter of the submacular hemorrhage needs to be less than 50% of the entire PED.
* Submacular fibrosis needs to be less than 50% of the entire PED.
* Sufficiently clear media (cornea, anterior chamber, lens, vitreous) for OCT, FA, and FP.
* Intraocular pressure of 25 mm or less in the study eye, with or without use of ocular hypotensive agents.

Exclusion Criteria:

* Pregnancy or lactation
* Premenopausal women not using adequate contraception
* Known serious allergies to ranibizumab, fluorescein dye, drug for pupillary dilation, topical anesthetic, sterilizing solution
* Contraindication to pupillary dilation in study eye
* Any condition (including inability to read visual acuity charts or language barrier) that may preclude patient's ability to comply with the study protocol requirements
* Presence of any advanced systemic condition or endstage disease, advanced Alzheimer syndrome, endstage cancer, etc., which will likely prevent patient from completing study.
* Previous therapeutic radiation in the region of the study eye.
* Prior anti-vascular endothelial factor therapy within 30 days.
* More than 3 sessions of prior anti-VEGF therapy.
* More than 1 prior photodynamic therapy (PDT)
* Prior triamcinolone in the past 6 months or dexamethasone in the past 1 month.
* Prior retinal pigment epithelial (RPE) tear in study eye.
* Prior ocular surgery (except YAG laser capsulotomy) for study eye within past 90 days.
* Anticipated ocular surgery (except YAG laser capsulotomy) for the next 12 months.
* Prior therapy for AMD (except minerals and vitamins), including laser, within the past 30 days.
* Prior intraocular or periocular corticosteroid therapy within the past 120 days
* Prior vitrectomy
* Presence of any causes of CNV and PED other than due to AMD.
* Presence of any substantial ocular disease (other than CNV and PED) that may compromise vision in the study eye and/or confound interpretation of the date; e.g. substantial cataracts, concomitant diabetic retinopathy affecting the macula, advanced glaucoma, optic neuritis, optic neuropathy or atrophy, marked macular atrophy, ocular vascular occlusion, history of retinal detachment, uveitis, viral or other forms of chorioretinitis, etc.
* Presence of ocular disease other than AMD affecting study eye, i.e. presumed ocular histoplasmosis syndrome, angioid streaks, pathologic myopia (spherical equivalent of greater than or equal to -8 diopters of myopia or axial length of greater than or equal to 25 mm), choroidal rupture, multifocal choroiditis, etc.
* Active ocular infection (i.e., bacterial, viral, parasitic, or fungal) in either eye at screening or Day 0.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-09; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Mean change in Best Corrected Visual Acuity from baseline measured at 4 meters on the ETDRS chart at 12 months. | 12 months

SECONDARY OUTCOMES:
Proportion of eyes reaching BCVA greater than or equal to 20/200 | 12 months
Proportion of eyes gaining greater than or equal to 0, 5, 10, and 15 letters on the ETDRS chart | 12 months
Reduction in central macular thickness from baseline (central 1-mm subfield) as measured by an OCT | 12 months
Changes in choroidal neovascular lesion (CNV)size on fluorescein angiography and fundus photography from baseline | 12 months
Changes in retinal pigment epithelial detachment size on fluorescein angiography and fundus photography, including height of the PED and associated submacular fluid on OCT in comparison to baseline | 12 months
Status of fluorescein staining or leakage (increased or decreased) from baseline | 12 months
Ocular safety outcome including ocular complication, i.e. RPE tears, uveitis, endophthalmitis | 12 months
Systemic safety outcome including cardiovascular event, cerebral vascular events | 12 months
Proportion of patients with an improvement from baseline in Contrast Sensitivity at 24 and 48 weeks | 24 and 48 weeks
Proportion of patients with an improvement from baseline in the VFQ overall composite score and near and distance activities subscales at 24 and 48 weeks | 24 and 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clement K Chan, M.D., Principal Investigator — Southern California Desert Retina Consultants
Locations (3):
- United States (3):
  - Jules Stein Eye Institute, Los Angeles, California
  - Southern California Desert Retina Consultants, Palm Desert, California
  - Black Hills Regional Eye Institute, Rapid City, South Dakota

REFERENCES:
- [Derived] Chan CK, Abraham P, Sarraf D, Nuthi AS, Lin SG, McCannel CA. Earlier therapeutic effects associated with high dose (2.0 mg) Ranibizumab for treatment of vascularized pigment epithelial detachments in age-related macular degeneration. Eye (Lond). 2015 Jan;29(1):80-7. doi: 10.1038/eye.2014.233. Epub 2014 Oct 3. PMID 25277305